CLINICAL TRIAL: NCT00797979
Title: Implant System for Fixation of Cranial Bone Flaps After Craniotomy for Brain Surgery
Acronym: CRANIOSG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080501
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Skull Fixation After Craniotomy for Neurosurgical Procedures
Keywords: Craniotomy; Skull fixation; Skull Grip; Reconstructive cranial surgery
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Skull Grip bone fixation
  Interventions: Device: Skull Grip bone fixation
- 2 (Active Comparator): Standard skull bon flap fixation, sutures
  Interventions: Device: sutures

INTERVENTIONS:
Device: Skull Grip bone fixation — Skull Grip bone fixation
  Arms: 1
Device: sutures — Standard skull bon flap fixation, sutures
  Other Names: Standard skull bon flap fixation, sutures
  Arms: 2

SUMMARY:
Bone flaps after craniotomy are typically fixed with suture material, mini plates and others devices. In some cases, fixation with suture material is not secure as it may result in shifting of the bone flap with its dislocation. We will test the safety and efficacy of SKULL GRIP a new device for fixation of the bone flap during cranial procedure comparing to traditional suture materials.

DETAILED DESCRIPTION:
At the end of the operation to start the fixation of cranial bone flaps, at least three Skull Grip titanium clamps will be positioned equidistant to one another along the craniotomy opening. The lower parts (complete circle) will be inserted between the dura and the cranium. The linear parts of the superior semicircle have to be in line with the craniotomy borders to allow the lodging of the bone flap. The different heights of the device are finalized to suit it for the different thickness of the cranial vault. The same procedure will be performed with all remaining Skull Grip titanium clamps.The bone flap will be then placed in its original position. By using a forceps, a simple and easy clockwise rotation of the superior semicircle will allow to block the SKULL GRIP clamp in place. For simple removal if necessary of the Skull Grip titanium clamps, even if bone ossification of the craniotomy edges has already occurred, it will be necessary just to lift up the superior semicircle of the Skull Grip by a forceps and to cut by a cutting forceps the pin between the two circle. Then, craniotomy could be completed in a standard way.

ELIGIBILITY:
Inclusion Criteria:

1. Major patient (aged ≥ 18 years)
2. Patient scheduled for craniotomy for a benign tumor
3. Patient informed and have signed informed consent

Exclusion Criteria:

1. Patient not affiliated with a social security scheme (or beneficiary entitled)
2. Patient with a known allergy to titanium
3. Patient non-compliant or whose follow-up to 3 months is impossible
4. Patient with against-indication scanner
5. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of the "Skull Grip" new system of cranial flap fixation | 2009

SECONDARY OUTCOMES:
To evaluate the security of "Skull Grip" new system of cranial flap fixation | 2009
Compare functional benefits (ease and speed of implementation) of "Skull Grip" new system of cranial flap fixation compared with traditional sutures | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore CHIBBARO, MD, Principal Investigator — Hôpital Lariboisière, Neurochirurgie
Locations (1):
- CHU Lariboisière, AP-HP, Neurochirurgie, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Chibbaro S, Makiese O, Bresson D, Hamdi S, Cornelius JF, Guichard JP, Reiss A, Bouazza S, Vicaut E, Ricci A, Galzio R, Poczos P, George B, Marsella M, Di Emidio P. Skull bone flap fixation - reliability and efficacy of a new grip-like titanium device (Skull Grip) versus traditional sutures: a clinical randomized trial. Minim Invasive Neurosurg. 2011 Oct;54(5-6):282-5. doi: 10.1055/s-0031-1297246. Epub 2012 Jan 25. PMID 22278799